CLINICAL TRIAL: NCT03449745
Title: Analysis of Immune Checkpoint Receptors Expression in the LIC Fraction pf AML Cells - ICAML-LIC
Brief Title: Immune Checkpoint Receptors in AML-Leukemic Initiating Cells
Acronym: ICAML-LIC
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2016/37
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; Immune Checkpoint Ligand; Flow Cytometry
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project aim at deciphering immune mechanisms that allow the immunoescape of AML initiating cells.

DETAILED DESCRIPTION:
Leukemic Initiating Cells (LIC) were shown to play a key role in AML relapses, and are characterized by resistance to treatment and a high capacity to escape to immune system. Immune checkpoints (ICP) maintain self-tolerance and physiological amplitude of the immune response. We decided to focus our work on ICP receptors and ligand that could be expressed by AML LIC and lymphocytes subsets. The tumor cells are able to express these ligands to exploit the ICP to overcome the anti-cancer immune response. Few studies are published in AML in the field of ICP, some studied limited cohort and others analyzed the expression of these ligands in total leukemic population, with a limited interest since the LIC fraction represents a small subset but mainly contributes to relapse. These cells are rare and their profile of expression could be highly different but not detectable in these studies because of technical limits. We aim at analyzing ICP ligands and receptors expression at diagnosis and relapse, the phenotype of BM cells will be analyzed by flow cytometry according to different panels of monoclonal antibodies using standard immunostaining protocols.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* newly diagnosed AML

Exclusion Criteria:

* isolated extramedullary AML
* mixed phenotype acute leukemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Acute Myeloid Leukemia
Sampling Method: Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2021-06-09 (Actual)

PRIMARY OUTCOMES:
Immune checkpoints (ICP) ligand expression | At inclusion
  Compare large panel of ICP ligand expression between LIC and HSC by flow cytometry

SECONDARY OUTCOMES:
Levels of ICP ligand expression | At inclusion
  Compare levels of ICP ligand expression according to FAB classification, cytogenetic classification and molecular abnormalities
Levels of ICP ligand expression | At inclusion
  Study levels of ICP ligand expression on minimal residual disease

CONTACTS AND LOCATIONS:
Overall Officials: Edouard FORCADE, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No